CLINICAL TRIAL: NCT03737266
Title: Sonographically Assisted Versus Conventionally Breast Surgery in Breast Cancer Patients With an Indication for Breast Conserving Surgery After Neoadjuvant Chemotherapy
Brief Title: Comparison of Conventional With Sonography Assisted Breast Surgery After Neoadjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Seno_Ex_MAC 003
Record Dates: First submitted 2018-10-16; First posted 2018-11-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonographically assisted breast surgery (Experimental): Sonography assisted breast surgery
  Interventions: Procedure: Sonographically assisted breast surgery; Procedure: Conventional breast surgery
- Conventional breast surgery (Active Comparator): Conventional breast surgery
  Interventions: Procedure: Sonographically assisted breast surgery; Procedure: Conventional breast surgery

INTERVENTIONS:
Procedure: Sonographically assisted breast surgery — Sonography
Procedure: Conventional breast surgery — Conventional

SUMMARY:
Aim of the study is to investigate whether intra-surgical visualisation of malignoma reduces the resection rate in the case of R1 resection compared to the procedure without sonographic visualisation

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years
* Female
* Presurgical validated breast cancer
* Unifocal to multifocal findings
* Palpable and/o non-palpable findings
* Neoadjuvant chemotherapy
* Indication for breast conserving therapy
* General operation ability and anesthesia ability
* Consent to conventional breast conserving breast surgery with wire marking
* Ability and will to follow the study conditions
* Written declaration of consent after clarification

Exclusion Criteria:

* Sonographically not clearly delineate resection areal
* Exclusion criteria for breast conserving therapy
* Simultaneous participation in other interventional trials that interfere with this study at the investigator's discretion

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 3 years
  proportion of surgical procedures for cancer in which the surgeon is able to completely remove all detectable tumor tissue with negative margins, indicating that no cancer cells remain in the surgical site

SECONDARY OUTCOMES:
Weight of primary resedate | 3 years
  weight of the tumor tissue removed during surgery for cancer
Time for cut and sew | During surgery
  duration of the surgical procedure from the initial incision to the completion of the closure of the incision site

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hahn, Prof. Dr., Principal Investigator — Department of Women's Health, University Hospital Tuebingen
Locations (1):
- Department for Women's Health, Tübingen, Baden-Wurttemberg, Germany